CLINICAL TRIAL: NCT06456905
Title: Automated Reinforcement Management Systems, Phase II
Acronym: ARMS II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington State University (Other)
Collaborators: Managed Health Connections (Unknown)
Responsible Party: Principal Investigator, Sterling McPherson, Principal Investigator, Washington State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19909
Record Dates: First submitted 2024-04-04; First posted 2024-06-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Alcohol Use Disorder
Keywords: alcohol consumption; contingency management; alcohol dependency; positive reinforcement; remote treatment; non-medicated assisted treatment; alcohol studies
MeSH Terms: conditions — Alcoholism; Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contingency Management + Treatment As Usual (Experimental): An experimental approach examining the effectiveness of contingency management for promoting a decrease in drinking through increasing rewards for positive behavior. Participants will be given positive reinforcement messaging regardless of the sample's results.
  Interventions: Behavioral: Contingency Management
- Non-Contingent Management + Treatment As Usual (No Intervention): Participants will be given a flat amount for submitting samples on time, and there is no increasing scale for maintaining samples at 0.00%BAC. Participants will be given positive reinforcement messaging regardless of the sample's results.

INTERVENTIONS:
Behavioral: Contingency Management — Participants in the contingent group will be rewarded on an incrementally increasing scale for submitting consecutive breathalyzer samples that are 0.00%. For every day this target is met, the participant will receive an increase in reward until a daily cap is reached. If a day contains at least one sample where the target is not met, the participant will not be paid for that day, and the amount will reset. The participant will have the opportunity to earn on this scale throughout the duration of the study.
  Arms: Contingency Management + Treatment As Usual

SUMMARY:
The Automated Reinforcement Management Systems Phase II (ARMS II) study is a phase II trial is a randomized controlled, non-medicated assisted trial to determine the effectiveness of Contingency Management (CM) treatment for reducing alcohol drinking among adults who want to quit or reduce their alcohol consumption.

DETAILED DESCRIPTION:
The Automated Reinforcement Management Systems Phase II (ARMS II) study is a phase II randomized controlled, non-medication assisted trial to determine the effectiveness of Contingency Management (CM) delivered remotely as a treatment for reducing alcohol consumption among drinking adults who want to reduce their consumption. The study will utilize an application developed by Managed Health Connections, Appropos Health, that connects to a Bluetooth breathalyzer to collect sample results and provide rewards to participants. Qualifying participants will be randomized into one of two groups, a Contingent or Non-Contingent group, and earn rewards based on the group they are randomized to. The contingent group will receive rewards on an escalating scale for submitting consecutive negative samples (0.00% BAC) at three time points per day: 11am, 4pm, and 9pm. The non-contingent group will earn rewards for submitting samples on time, independent of the test results. All rewards will be given in the form of electronic vouchers, which can be exchanged for a merchant of the participant's choosing. All participants will be invited to complete short, daily surveys, and will be called once per week by a research coordinator for a check in on the study's progress. All participants will be invited to the research clinic once per month. All participants will additionally receive positive messaging to reinforce positive behavior, or provide support to encourage a change in behavior.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years
* Have consumed 3 or more drinks in once occasion 4 or more times in the previous 30 days 3
* Have the ability to read and speak English
* Have the ability to provide written informed consent
* Have a breath alcohol value of 0.00 during informed consent
* Owns a smartphone with an active service provider that is compatible with the study application.

Exclusion Criteria:

* Severe alcohol use disorder that our medical staff deems too risky for safe participation;
* Significant risk of dangerous alcohol withdrawal, defined as history of seizure due to alcohol withdrawal in the last 12 months and/or expression of concern by the participant about dangerous withdrawal
* Anyone aged 71 or older.
* Anyone with a suicide attempt in the last 2 years.
* Individuals who express concern regarding dangerous withdrawal or who exhibit dangerous withdrawal symptoms.
* Individuals who do not test BrAC = 0.00 on the breathalyzer during the baseline visit.
* Any other condition that investigators determine a medical or psychiatric condition that would compromise safe study participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2024-06-07 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in days abstinent | 45 months
  Increase in days abstinent as verified through three consecutive negative breathalyzer samples submitted at designated time slots over a period of 12 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Sterling M McPherson, PhD, Principal Investigator — Washington State University
Locations (1):
- Washington State University, Spokane, Washington, United States